CLINICAL TRIAL: NCT05870878
Title: Generation R Next - Optimaal Opgroeien
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: INDIGO Rijnmond (Unknown); ZonMw: The Netherlands Organisation for Health Research and Development (Other); Stichting Bevordering van Volkskracht (Unknown); Stichting Achmea Gezondheidszor (Other); Bernard van Leer Foundation (Unknown); Ministerie van Volksgezondheid, Welzijn en Sport (Unknown)
Responsible Party: Principal Investigator, Vincent Jaddoe, Prof. dr., Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MEC-2022-0440, NL81446.078.22
Record Dates: First submitted 2023-03-25; First posted 2023-05-23 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Pregnancy Early; Outcome, Adverse Birth; Lifestyle Factors; Preconception Care; Pregnancy Outcome; Pregnancy Complications; Risk Reduction Behavior
MeSH Terms: conditions — Pregnancy Complications; Risk Reduction Behavior | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Block randomisation with stratification factor: pregnancy status (yes/no)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard care and additional lifestyle program (Experimental): 3 lifestyle group sessions (1 physical and 2 online) and additional online platform and individual consultation given at the research center by trained employees
  Interventions: Other: Standard care; Other: Lifestyle program
- Standard care (Other): Individual consultation given at the research center by trained employees
  Interventions: Other: Standard care

INTERVENTIONS:
Other: Standard care — Individual lifestyle consultation
Other: Lifestyle program — Lifestyle program focusing on lifestyle advice, coping with stress and adherence to a healthy(er) lifestyle. This program consists of 3 group sessions and an online platform.
  Arms: Standard care and additional lifestyle program

SUMMARY:
The aim of this randomized controlled trial is to improve birth outcomes and long-term outcomes in mother and child by optimizing lifestyle,nutrition and stress experience in the preconception period and early pregnancy in women and men

The main research question that will be addressed is: Does an intervention focused on optimizing preconception and early pregnancy lifestyle, nutrition and stress improve the birth outcomes and long-term outcomes in mother and child?

Participants will receive an individual lifestyle consultation at the start of the study. Depending on their study arm, participants will receive an additional lifestyle program focused on health during preconception and early pregnancy, coping with stress and adherence to a healthy(er) lifestyle. The given advices are based on national guidelines.

Researchers will compare the intervention group and control group to see if (adherence to) this lifestyle program improve birth outcomes and long-term outcomes in mother and child.

DETAILED DESCRIPTION:
Preconception and early pregnancy are critical periods for health and wellbeing across the full life course in the offspring. Improving lifestyle, nutrition and stress in both women and their partners already from the preconception period onwards may have beneficial effects on the offspring.

This RCT will include preconception/early pregnancy integrated life style intervention focused on a healthy weight (BMI: 18.5-25 kg/m2), stopping alcohol/smoking/drugs, supplementing folic acid and vitamin D, a healthy diet (weekly fish, iron and vitamin C rich food) and stress reduction. Reducing stress appears to be effective for improving (maternal) health and reducing risk behavior. Mind-body therapy, a combination of yoga exercises and mindfulness seems to be a popular intervention, especially among pregnant women or women of childbearing age from various ethnic backgrounds.

The use of the preconception consultation is not yet optimal. This is partly due to the difficulty of reaching (vulnerable) groups and the limited insight regarding the efficacy.

The aim of this randomized controlled trial is to improve birth outcomes and long-term outcomes in mother and child by optimizing lifestyle in the preconception period and early pregnancy in women and men. The main research question is whether an intervention focused on optimizing preconception and early pregnancy lifestyle, nutrition and stress improves the birth outcomes and long-term outcomes in mother and child?

This RCT will be embedded in the available Generation R Next research infrastructure.

Prior to randomization, the intervention and control groups will be offered an individual lifestyle consultation for both women and men, and, if pregnant, an early pregnancy ultrasound. After randomization, there will be two groups: the intervention group and the control group. Both groups will receive standard care, including an individual lifestyle consultation in line with current national standards for preconception and early pregnancy. The intervention group will additionally attend three group sessions (online and physical) focused on health during preconception and early pregnancy, coping with stress and adherence to a healthy lifestyle. The advices are based on national guidelines for health during the preconception period and early pregnancy. Compliance with the prescribed advice is encouraged via newly developed digital platform

ELIGIBILITY:
Inclusion Criteria:

Women and their parents:

* Planning a pregnancy or early pregnancy up to < 12 weeks
* With the presence of at least one of the predetermined risk factors
* Residential address in the municipality of Rotterdam and expected residential address in the municipality of Rotterdam at the birth of their child
* Consent for participation

Exclusion Criteria:

Women and their partners:

* Temporary or complete withdrawal from participation
* Gestational age > 12+0 at study entry

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1750 (Estimated)
Dates: Start 2023-01-19 (Actual); Primary Completion 2026-05-08 (Estimated); Study Completion 2030-11-08 (Estimated)

PRIMARY OUTCOMES:
Preterm birth | Assessed at birth
  Birth of the child before 37 weeks of pregnancy
Low birthweight/small-for-gestational-age | Assessed at birth
  Birthweight below 10th percentile corrected for gestational age
High birthweight/large-for-gestational-age | Assessed at birth
  Birthweight above 90th percentile corrected for gestational age
Low Apgar-score | Assessed at birth
  Apgar-score assessed 5 minutes after birth, below 7 is considered as low with higher chance on worse outcome (scale: 0-10)
Birth weight | Assessed at birth
  Birth weight measured continuously

SECONDARY OUTCOMES:
Adherence to lifestyle advice (mother) | During pregnancy and early childhood, until 12 months
  Lifestyle changes assessed via questionnaires during the study period
Sleep/wake rhythm (mother) | During pregnancy and early childhood, until 12 months
  Sleep/wake rhythm assessed via questionnaires during the study period with the Munich Chronotype Questionnaire (MCTQ). 12 items
Sleep/wake rhythm (mother) | During pregnancy and early childhood, until 12 months
  Sleep/wake rhythm assessed via questionnaires during the study period with the General Sleep Disturbances Questionnaire. 22 items, responses are given on an eight-point scale ranging from 0 (no days) to 7 (every day). The total score for the scale ranges between 0 and 154, with higher scores indicating a higher frequency of sleep disturbances.
Social support (mother) | During pregnancy and early childhood, until 12 months
  Social support assessed via questionnaires during the study period with the Adaptive Functioning Scales Spouse/Partner. 6 items with 6-point Likert scale.
Experience of stress (mother) | During pregnancy and early childhood, until 12 months
  Experience of stress assessed via questionnaires during the study period with the brief symptom inventory (BSI). 53 items with 5-point Likert scale.
Weight gain during pregnancy (mother) | During pregnancy and early childhood, until 12 months
  Weight gain during pregnancy assessed via questionnaires during the study period and with weight measurements during the pregnancy visits at the research center measured in kilogram
Weight maintenance after 6 and 12 months pregnancy (mother) | 12 months after birth of the child
  Weight maintenance after 6 and 12 months of pregnancy assessed via questionnaires during the study period
Time to pregnancy (mother) | At delivery
  Time to pregnancy assessed via questionnaires regarding menstrual period and conception during the study period
Occurrence of miscarriage (mother) | At delivery
  Occurrence of miscarriage assessed via questionnaires during the study period
Glucose metabolism and diabetes during pregnancy (mother) | At delivery
  Glucose metabolism assessed via taken blood samples (measured: glucose in mmol/L, normal range: 4-8 mmol/L) at visits in first trimester and 30 weeks of pregnancy
Occurrence of gestational hypertensive disorders during pregnancy (mother) | At delivery
  Occurrence of gestational hypertensive disorders assessed via questionnaires during the study period and with blood pressure measurements during the pregnancy visits at the research center measured in systolic and diastolic millimetre of mercury (mmHg). Cutoff values: 140 systolic and 80 diastolic.
Adherence to lifestyle advice (partner) | During pregnancy and early childhood, until 12 months
  Lifestyle changes assessed via questionnaires during the study period
Sleep/wake rhythm (partner) | During pregnancy and early childhood, until 12 months
  Sleep/wake rhythm assessed via questionnaires during the study period with the Munich Chronotype Questionnaire (MCTQ). 12 items
Sleep/wake rhythm (partner) | During pregnancy and early childhood, until 12 months
  Sleep/wake rhythm assessed via questionnaires during the study period with the General Sleep Disturbances Questionnaire. 22 items, responses are given on an eight-point scale ranging from 0 (no days) to 7 (every day). The total score for the scale ranges between 0 and 154, with higher scores indicating a higher frequency of sleep disturbances.
Social support (partner) | During pregnancy and early childhood, until 12 months
  Social support assessed via questionnaires during the study period with the Adaptive Functioning Scales Spouse/Partner. 6 items with 6-point Likert scale.
Experience of stress (partner) | During pregnancy and early childhood, until 12 months
  Experience of stress assessed via questionnaires during the study period with the brief symptom inventory (BSI). 53 items with 5-point Likert scale.
Growth and adiposity (child) | 1, 3, 6 and 12 months of age
  Growth of the child assessed via questionnaires during the study period and via weight and height measurements at the consultation office (unit: kilograms and centimeters)
Development and behavior (child) | 1, 3, 6 and 12 months of age
  Development and behavior of the child assessed via questionnaires during the study period (Child Development Inventory. 30 items) and via behavioral assessment at the consultation office.
Overall health (child) | 1, 6 and 12 months of age
  Overall health of the child assessed via questionnaires during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Jaddoe, Prof.dr., Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No